CLINICAL TRIAL: NCT03078218
Title: Health-economic Impact of Pulse Oximetry Systematic Screening of Critical Congenital Heart Disease in Asymptomatic Newborns
Acronym: OXYNAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2015/27
Record Dates: First submitted 2017-02-06; First posted 2017-03-13 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Critical Congenital Heart Disease
Keywords: Pulse oximetry; Asymptomatic newborns
MeSH Terms: interventions — Oximetry

STUDY DESIGN:
Intervention Model Description: Multicenter controlled before and after study conducted in Nouvelle Aquitaine, including types 1, 2 and 3 maternity wards.
  The BEFORE period will be strictly observational in order to assess the current screening strategy as it is conducted in real life.
  The AFTER period will be consist in a systematic pulse oximetry screening where all eligible newborns will be included in the same maternity wards as the BEFORE period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before period group (No Intervention): Strictly observational in order to assess the current screening strategy as it is conducted in real life
- After period group (Experimental): Consist in a systematic pulse oximetry screening where all eligible newborns will be included in the same maternity wards
  Interventions: Diagnostic Test: Pulse oximetry

INTERVENTIONS:
Diagnostic Test: Pulse oximetry — The tool evaluated will be the assumption of peripherical arterial oxygen saturation by pulse oximetry. The pulse oximetry will identify hypoxemic CCHD and hypoxemic non-cardiac disease before discharge.The test will be realised before 24 hours of life in a newborn aged at least of 35 weeks of gestation.
  Arms: After period group

SUMMARY:
Persistant hypoxemia in the newborn confers, even isolated, an abnormal clinical situation, that needs to be addressed for an adequate diagnosis and an optimal treatment.

If during the first hours of life, hypoxemia is frequent and often transient, beyond that, it is necessary to search the various etiological conditions such as a critical congenital heart disease (CCHD) or a non cardiac affection (sepsis, anemia, respiratory disease).

Newborn pulse oximetry screening identifies babies with critical congenital heart disease (CCHD) based on the rational that they frequently have a degree of hypoxemia that may be clinically undetectable. CCHDs are life-threatening forms of congenital heart disease (CHD) occuring in 2-3/1000 live births but accounting for 3%-7.5% of infant deaths.

Early detection is beneficial because of acute collapse, if not resulting in death, is associated with a worse surgical and neurodevelopmental outcome.

Currently, screening for CCHD involves antenatal ultrasound scanning and post-natal physical examination. Although antenatal detection rates have improved over recent years and can be as high as 70%-80% in some centers, this is not consistent. Indeed, in "Nouvelle Aquitaine" overall <50% of CCHDs are detected before birth. In addition, up to a third of infants with CCHD may be missed on post-natal examination. Pulse oximetry screening can help to close the "diagnostic gap' that is, increase the detection of babies who slip through the current screening net.

Several large European studies and a subsequent meta-analysis have shown that pulse oximetry screening is a highly specific (99.9%) and moderately sensitive (76.5%) test which increases CCHD detection rates. The high specificity results in a low false-positive rate 0.05% to 0.5%. But those babies with a Positive Test, if they may not have CCHD, they may be diagnosed with other causes of hypoxemia (congenital pneumonia, sepsis, persistent pulmonary hypertension,...). As with CCHD, delayed recognition of these conditions can result in postnatal collapse and significant morbidity and mortality. It is also more useful to consider these conditions as secondary targets of screening and to remember they constitute 30%-70% of false positives. In 2011, the US Health and Human Services Secretary recommended that pulse oximetry screening for CCHD be added to the Recommended Uniform Screening Panel. In Europe, implementation is advanced in such countries as North European Countries, and Switzerland. There isn't yet any European guidance. In France, the implementation is limited to local and transient experiments. The feasibility, usefulness and cost-effectiveness of routine pulse oximetry screening have not been evaluated so far. The French setting has two specificities : 1/ the antenatal detection rate is considered to be rather high. 2/ in contrast to a lot of other European countries, early discharge from the maternity ward before 48 hours of life is not common, decreasing the risk of discharging a baby with undiagnosed CCHD, but not saving babies from collapse.

- The Investigators hypothesis is that routine pulse oximetry screening in asymptomatic newborns would allow to reduce the incidence of complications related to CCHDs as well as those related to non cardiac pathologies for a reasonable cost for the French Health Care System.

ELIGIBILITY:
Inclusion Criteria:

BEFORE Period: newborns

* aged at birth superior or equal to 35 weeks of gestation (≥ 35+ 0 days weeks of gestation)
* borned in metropolitan France in involved maternity wards.
* Asymptomatic before the screening (no respiratory signs, neither collapse or cardiac arrest).

AFTER Period: newborns

* aged at birth superior or equal to 35 weeks of gestation (≥ 35+ 0 days weeks of gestation)
* borned in metropolitan France in involved maternity wards.
* Asymptomatic before the screening (no respiratory signs, neither collapse or cardiac arrest).
* With consent done by the 2 parents.
* Parents covered with the French National health insurance

Exclusion Criteria:

* Newborns with a prenatally diagnosed congenital cyanotic malformation or any other cyanotic affection.
* Newborns with a postnatal pre-screening diagnosed congenital cyanotic malformation or any other cyanotic affection.

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44140 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Incremental cost-effectiveness ratio | Up to 12 month of each period
  Difference of mean costs between the two strategies divided by the difference in the number of complications between the two strategies. Complications of interest are: acute respiratory distress, acute cardio-circulatory distress (collapse, acidosis, shock, multivisceral failure), and death.

SECONDARY OUTCOMES:
Incremental cost per life saved | Up to 12 month of each period
  Difference of mean costs between the two strategies divided by the difference in the number of saved lives between the two strategies.
Net monetary benefit for the French Health System of generalizing the pulse oximetry screening | Up to 12 month of each period
Cost of pulse oximetry screening for critical congenital heart defects in France. | The duration of a pulse oximetry examination
  Costs will be calculated in the perspective of the French Health System. The test will be realised before 24 hours of life in a newborn aged at least of 35 weeks of gestation
Performances of pulse oximetry for the diagnostic of CCHD and non-cardiac disease | Up to 12 month of the after period
  sensibility, specificity, positive predictive value, negative predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Julie THOMAS, MD, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux
Locations (29):
- France (29):
  - CH Agen, Agen
  - Clinique Esquirol - Saint Hilaire, Agen
  - CH Angoulême, Angoulême
  - CH de la Haute Gironde, Blaye
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH Brive, Brive-la-Gaillarde
  - Clinique Jean Villar, Bruges
  - CH Châtellerault, Châtellerault
  - CH Dax, Dax
  - CH Guéret, Guéret
  - Maternité Pernelle d'Aufrédy CH de La Rochelle - Ré - Aunis, La Rochelle
  - CH d'Arcachon, La Teste-de-Buch
  - CH Robert Boulin, Libourne
  - CHU Limoges, Limoges
  - Clinique Emailleurs, Limoges
  - Polyclinique Rive droite, Lormont
  - CH Marmande, Marmande
  - CH Mont de Marsan, Mont-de-Marsan
  - CH Niort, Niort
  - CHU de Bordeaux, Pessac
  - CH Périgueux, Périgueux
  - CHU de Poitiers, Poitiers
  - CH Rochefort, Rochefort
  - CH Saint Junien, Saint-Junien
  - CH Saintes, Saintes
  - Clinique Soyaux, Soyaux
  - Maison de Santé Protestante de Bordeaux Bagatelle, Talence
  - CH de Tulle, Tulle
  - CH Villeneuve-sur-Lot, Villeneuve-sur-Lot

IPD SHARING:
Plan to Share IPD: No